CLINICAL TRIAL: NCT02447146
Title: Effects of Resistance Training on Bradykinesia and Physical Function in Patients With Parkinson's Disease.
Brief Title: Resistance Training in Patients With Parkinson's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Wagner Rodrigues Martins, Professor, University of Brasilia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RT-PD
Record Dates: First submitted 2015-05-12; First posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training group (Experimental): 9-week resistance training program
  Interventions: Other: Resistance Training
- Control group (Other): 'Lectures on the disease'
  Interventions: Other: Lectures on the disease

INTERVENTIONS:
Other: Resistance Training — The TG performed the RT program using weight machines. Before the training period, participants underwent three weeks with eight familiarization sessions to ensure proper technique execution. The protocol aimed to workout major muscle groups and involved the following exercises: chest press, knee extension, hamstrings curl, leg press, and seated row. Training sessions lasted approximately 50-60 minutes with 2 sets of 10-12 repetitions until fatigue.
  Arms: Training group
Other: Lectures on the disease — The control group attended an orientation program with lectures on health, quality of life and scientific update on disease.
  Arms: Control group

SUMMARY:
This is a controlled trial to assess the effects of resistance training on bradykinesia and physical function in patients with Parkinson's Disease. Forty patients diagnosed with Parkinson Disease stage 1 to 3 of the Hoehn and Yahr scale took part in the study and were allocated into 2 groups; Training Group performed a 9-week RT program twice a week while the Control Group attended lectures on the disease.

ELIGIBILITY:
Inclusion Criteria:

* Medical neurologist confirmation of 1-3 Hoehn and Yahr stages,
* age between 50 and 80 years old;
* and physician attested to participate in the resistance training program.

Exclusion Criteria:

* Diagnostic of any other neurological disease, cardiovascular disease, hematologic or orthopedic disorders;
* and motor fluctuations or severe dyskinesia that could affect their ability to perform the experimental protocol.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Bradykinesia measured with Unified Parkinson's Disease Rating Scale, section III | One time point; after the end of 9-week resistance training
Functional Performance measured with Ten Meters Walk Test. | One time point; after the end of 9-week resistance training

SECONDARY OUTCOMES:
Muscle strength measured with isokinetic peak torque. | One time point; after the end of 9-week resistance training

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Oliveira, PhD, Study Director — College of Physical Education - University of Brasilia

REFERENCES:
- [Background] Dibble LE, Hale TF, Marcus RL, Droge J, Gerber JP, LaStayo PC. High-intensity resistance training amplifies muscle hypertrophy and functional gains in persons with Parkinson's disease. Mov Disord. 2006 Sep;21(9):1444-52. doi: 10.1002/mds.20997. PMID 16773643
- [Background] Falvo MJ, Sirevaag EJ, Rohrbaugh JW, Earhart GM. Resistance training induces supraspinal adaptations: evidence from movement-related cortical potentials. Eur J Appl Physiol. 2010 Jul;109(5):923-33. doi: 10.1007/s00421-010-1432-8. Epub 2010 Mar 21. PMID 20306270
- [Background] Fisher BE, Wu AD, Salem GJ, Song J, Lin CH, Yip J, Cen S, Gordon J, Jakowec M, Petzinger G. The effect of exercise training in improving motor performance and corticomotor excitability in people with early Parkinson's disease. Arch Phys Med Rehabil. 2008 Jul;89(7):1221-9. doi: 10.1016/j.apmr.2008.01.013. Epub 2008 Jun 13. PMID 18534554
- [Result] Allen NE, Canning CG, Sherrington C, Fung VS. Bradykinesia, muscle weakness and reduced muscle power in Parkinson's disease. Mov Disord. 2009 Jul 15;24(9):1344-51. doi: 10.1002/mds.22609. PMID 19425085